CLINICAL TRIAL: NCT05590299
Title: A Randomised, Controlled Trial Evaluating the Effectiveness of Fish Oral Immunotherapy (FOIT) in Inducing Desensitisation or Remission in Children With Fish Allergy Compared With Placebo
Brief Title: Fish Oral Immunotherapy in Hong Kong Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Agnes Sze-Yin Leung, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FOIT
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Fish Allergy; Food Allergy in Children
Keywords: Fish allergy; Codfish; Oral immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish oral immunotherapy (Active Comparator): Fish oral immunotherapy to be taken daily for 12 months.
  Interventions: Other: Fish oral immunotherapy (codfish)
- Placebo (Placebo Comparator): Placebo oral immunotherapy to be taken daily for 12 months.
  Interventions: Other: Placebo oral immunotherapy

INTERVENTIONS:
Other: Fish oral immunotherapy (codfish) — Codfish in mixture of potato prepared under food manufacturing regulations provided in varying doses
  Arms: Fish oral immunotherapy
Other: Placebo oral immunotherapy — Placebo in potato mixture prepared under food manufacturing regulations provided in varying doses
  Arms: Placebo

SUMMARY:
At present there is no cure for food allergy. People with a food allergy need to avoid the food they are allergic to in order to stay safe, but we know that accidental exposure is common. Researchers have begun to look at the effectiveness of 'oral immunotherapy' as a treatment for food allergy but results have been mixed.

This study is a randomized controlled trial to evaluate the effectiveness of Fish Immunotherapy (FOIT), with codfish as the primary focus, in inducing tolerance in children with fish allergy compared with Placebo. Children will take increasing doses of codfish protein until a total of 12 months treatment is completed. Children will be tested for fish allergy at the start of the study, at the end of fish treatment T1 (12 months) and T2 (8 weeks) after treatment.

DETAILED DESCRIPTION:
This is a two-armed, randomised (1:1), blinded, placebo-controlled, parallel-group, superiority trial.

The study consists of:

Screening visit occurs within three months before Day 1.

Day 1 Rush Induction Phase is the start of treatment where participants receive increasing doses of fish (or placebo) OIT every 20 minutes to reach a predefined dose of fish protein (or placebo).

Week 1 - 12 is the Buildup Phase where the daily dose of fish (or placebo) OIT is increased every 2 weeks* until a maintenance dose of fish protein (or placebo) is reached. This is expected to take 12 weeks.

Week 13 - 52 is the Maintenance Phase where participants take a daily dose of fish protein (or placebo) at home and continue until a total of 12 months of treatment is completed.

Week 53 - 59 is the Elimination Phase where participants continue on a fish-elimination diet post-treatment.

The primary outcome analysis will be conducted when all subjects have either completed the T2 DBPCFC or terminated the study prior to their T2 visit. Analysis of safety and tolerability, and other secondary outcomes to the T2 timepoint will also be conducted at this time.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 2 year and 10 years of age
* >7kg (the weight considered safe for the administration of an adrenaline autoinjector) (e.g. Jext)
* Confirmed diagnosis of codfish allergy as defined by a failed DBPCFC with codfish and a positive SPT (>=3mm than control) or sIgE to codfish (of at least 0.35 kUA) at screening.

Exclusion Criteria:

* Serum codfish-specific IgE antibody level > 100 kUA/L
* History of severe anaphylaxis (as defined by persistent hypotension, collapse, loss of consciousness, persistent hypoxia or ever needing more than three (3) doses of intramuscular adrenaline or an intravenous adrenaline infusion for management of an allergic reaction)
* Severe anaphylaxis during the study entry DBPCFC (defined as persistent hypotension, collapse, loss of consciousness, persistent hypoxia, or requiring more than 3 doses of intramuscular adrenaline or an intravenous adrenaline infusion for management of an allergic reaction)
* FEV1 <85% at rest and FEV1/FVC ≤ 85% at rest or ongoing chronic persistent asthma (as per Australian Asthma Foundation guidelines)
* Underlying medical conditions (e.g. cardiac disease) that increase the risks associated with anaphylaxis
* Use of beta-blockers, and ACE inhibitors
* Inflammatory intestinal conditions, indwelling catheters, gastrostomies, immune-compromised states, post-cardiac and/or gastrointestinal tract surgery, critically-ill and those requiring prolonged hospitalisation or other conditions that may increase the risks of probiotic associated sepsis
* Reacting to the placebo component during the study entry DBPCFC
* Have received other food immunotherapy treatment in the preceding 12 months
* Currently taking immunomodulatory therapy (including allergen immunotherapy)
* Past or current major illness that in the opinion of the Site Investigator may affect the subject's ability to participate in the study e.g. increased risk to the participant
* History of suspected or biopsy-confirmed eosinophilic oesophagitis (EoE)
* Subjects who in the opinion of the Site Investigator are unable to follow the protocol

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve full desensitisation (passed T1 challenge) in OIT vs placebo. | T1 - One Day after final day of maintenance treatment

SECONDARY OUTCOMES:
Proportion of participants with 8-week sustained unresponsiveness (passed T1 and T2 challenges) in OIT vs placebo. | T2 - 8 weeks after final day of maintenance treatment
The cumulative dose tolerated during the T1 challenge in OIT vs placebo. | T1 - One Day after final day of maintenance treatment
Skin prick test wheal size and fish-specific IgE to fish in OIT vs placebo. | M1 - At 6 months of treatment; T1 - One Day after final day of maintenance treatment. T2 - 8 weeks after final day of maintenance treatment
Exposure-adjusted incidence rate and severity of treatment emergent adverse events (TEAEs) in OIT vs placebo. | TEAEs will be collected until T2 - 8 weeks after final day of maintenance

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study information — https://www.allergycuhk.org/foit